CLINICAL TRIAL: NCT02516657
Title: Effect of Liraglutide on Glycemic Control, Glucagon Secretion and Inflammatory Markers in Adolescents With Type 1 Diabetes Mellitus
Brief Title: Liraglutide in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Lucy D. Mastrandrea, Associate Professor, University at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 437619-6
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Liraglutide 0.6 mg (Experimental): Liraglutide 0.6 mg daily injection x 7 days
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide 0.6 mg
  Other Names: Victoza

SUMMARY:
The purpose of this study is to study the effect of a liraglutide, a glucagon-like peptide agonist, on post-meal blood glucose concentrations, glucagon levels, mean weekly blood sugars, and insulin doses in adolescents with Type 1 diabetes. Type 1 diabetes is an autoimmune disease that is usually diagnosed before the age of 20. Individuals with this disease are completely dependent on insulin for survival. While significant advances have been made in technological support for improving diabetes control, insulin remains the only effective treatment for Type 1 diabetes. Liraglutide is a long-acting glucagon-like peptide-1 analog. This drug is approved for the treatment of Type 2 diabetes in adults. This study will test the effect of liraglutide on blood sugar control in adolescents with Type 1 diabetes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1DM) affects approximately 1:500 children and represents the major form of diabetes in the pediatric population (1). Diagnosis of T1DM is based on symptoms consistent with hyperglycemia (polyuria, polydipsia, and weight loss) and elevated blood sugars. Diagnosis of T1DM is confirmed by measuring serum autoantibodies against insulin and other beta-cell proteins. Subcutaneous insulin is the mainstay of diabetes care; however, ability to achieve optimal glycemic control is impacted by multiple factors including diet, exercise, and psychosocial barriers.

The Diabetes Control and Complications Trial and follow-up EDIC trial were landmark studies demonstrating that improving glycemic control significantly reduces the risk of both micro and macro-vascular disease (2). While technologic advances in blood sugar monitoring, insulin analogs and insulin delivery devices have been made, it is estimated that less than 40% of individuals meet recommended glycemic standards as set forth by the American Diabetes Association; these estimates may be lower in the pediatric population. Thus, adjuvant pharmacologic therapies that improve glycemic control are being tested in patients with T1DM.

Incretin hormones are a class of intestinal peptides that are released in response to nutrient intake (3). The best described incretin hormones are glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP). These hormones act at the level of direct stimulation of pancreatic β-cell function and through extra-pancreatic mechanisms. They primarily potentiate glucose-dependent insulin secretion from the β-cell; other β-cell effects include increasing insulin biosynthesis, stimulating β-cell replication, and preventing apoptosis. Secondary effects of incretin hormones include suppression of glucagon secretion, inhibition of gastric emptying, and potentiation of hepatic glucose uptake (3).

Currently, there are two GLP-1 analogs approved by the Food and Drug Adminstration as adjuvant treatment of Type 2 diabetes mellitus in adults (> 18 years) who fail to reach glycemic targets with metformin and/or oral hypoglycemic agents. The two drugs - exenatide (BID) and liraglutide (QD) are administered subcutaneously. They have been demonstrated to improve glycemic control in this population and, in some individuals, lead to sustained weight loss.

This study aims to determine whether acute exposure to liraglutide decreases the mean weekly blood glucose levels in adolescents with T1DM. In addition, we will determine whether liraglutide decreases glucose excursions following a meal challenge. The overall hypothesis to be tested is that short-term exposure (7 days) to liraglutide improves glycemic control in adolescents/young adults with T1DM treated with continuous subcutaneous insulin infusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus greater than 1 year
* Insulin regimen - continuous subcutaneous insulin infusion with continuous glucose monitoring device
* HbA1c <10%

Exclusion Criteria:

* Previous exposure to liraglutide
* History of abdominal surgery
* Gastrointestinal reflux disease
* History of acute or chronic pancreatitis
* History of alcohol abuse or unwillingness to abstain from alcohol during the study
* History of thyroid cancer
* Family history of Multiple Endocrine Neoplasia 2B syndrome
* Pregnant/breastfeeding females
* Individuals with antibody-negative insulin requiring diabetes that is consistent with Monogenic Diabetes of Youth
* Individuals with steroid induced or cystic fibrosis related diabetes

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy D Mastrandrea, MD, PhD, Principal Investigator — University at Buffalo
Locations (1):
- UBMD Pediatrics, Division of Pediatric Endocrinology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from medical clinic
Period: Overall Study
Arm/Group | Liraglutide 0.6 mg
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 5 adolescents with Type 1 diabetes for > 1 year
Arm/Group | Liraglutide 0.6 mg
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent of glycosylated HemoglobinA] — Hemoglobin A1c for participants at baseline visit
  Percent of glycosylated HemoglobinA | 8.52 (0.64)
Total Daily insulin dose [Mean (Standard Deviation); unit: Units per day] | 73.74 (10.09)

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Blood Glucose
Description: The primary outcome is to determine whether liraglutide decreases mean weekly blood glucose (mean mg/dL glucose as measured by continuous glucose monitor readings) in adolescents with Type 1 diabetes
Time Frame: Visit 1 (Before Liraglutide) at baseline (Day 0) vs. Visit 2 (After Liraglutide) on Day 7;
Population: Data for mean weekly blood glucose was only collected for 4 of the 5 subjects enrolled in the study. 1 subject had missing CGM data
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Liraglutide 0.6 mg
Number analyzed (Participants) | 4
mg/dL
  Visit 1, before liraglutide | 187 (35)
  Visit 2, after liraglutide | 178 (42)

2. Secondary Outcome: Total Daily Insulin Dose
Description: mean U/kg/day over 7 days
Time Frame: Visit 1 (Before Liraglutide) at baseline (Day 0) vs. Visit 2 (After Liraglutide) on Day 7;
Population: Unable to determine mean U/kg/day for one of the subjects due to missing data
Measure: Mean (Standard Deviation); unit: U/kg/day
Groups:
- Before Liraglutide: U/Kg/Day before liraglutide administered
- Liraglutide Treatment: U/kg/day during liraglutide treatment
Arm/Group | Before Liraglutide | Liraglutide Treatment
Number analyzed (Participants) | 4 | 4
U/kg/day | 0.97 (0.18) | 0.67 (0.14)

3. Other Pre Specified Outcome: Blood Sugar < 70 mg/dL
Description: Determine whether liraglutide increases episodes of blood sugar <70 mg/dL as measured by glucometer and CGM
Time Frame: Visit 1 (Before Liraglutide) at baseline (Day 0) vs. Visit 2 (After Liraglutide) on Day 7;
Population: Unable to determine mean U/kg/day for one of the subjects due to missing data
Measure: Mean (Standard Deviation); unit: episodes
Groups:
- Before Liraglutide: BS < 70 mg/dL before liraglutide
- Liraglutide Treatment: BS <70 mg/dL during liraglutide treatment
Arm/Group | Before Liraglutide | Liraglutide Treatment
Number analyzed (Participants) | 4 | 4
episodes | 5.5 (7.7) | 3.3 (3.3)

4. Other Pre Specified Outcome: Serum Amylase Level
Description: Determine amylase levels before and during liraglutide treatment
Time Frame: Visit 1 (Before Liraglutide) at baseline (Day 0) vs. Visit 2 (After Liraglutide) on Day 7;
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Before Liraglutide: Amylase before liraglutide
- Liraglutide Treatment: Amylase during liraglutide treatment
Arm/Group | Before Liraglutide | Liraglutide Treatment
Number analyzed (Participants) | 5 | 5
U/L | 36 (15) | 33 (11)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Liraglutide 0.6 mg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT02516657/Prot_SAP_000.pdf